CLINICAL TRIAL: NCT04151680
Title: Safety and Efficacy of Anticoagulation on Demand After Percutaneous Coronary Intervention in High Bleeding Risk (HBR) Patients With History of Paroxysmal Atrial Fibrillation
Brief Title: Anticoagulation on Demand After Percutaneous Coronary Intervention in High Bleeding Risk Patients
Acronym: INTERMITTENT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Professor, University of Roma La Sapienza
Other Study IDs: 2019/D/983
Record Dates: First submitted 2019-10-30; First posted 2019-11-05 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Ischemic Heart Disease; Atrial Fibrillation
Keywords: coronary artery disease
MeSH Terms: conditions — Myocardial Ischemia; Atrial Fibrillation; Coronary Artery Disease | interventions — Rivaroxaban; apixaban; edoxaban

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intermittent anticoagulation: Patients receiving anticoagulation only if continuous electrocardiographic monitoring detects an atrial fibrillation episode
  Interventions: Drug: Intermittent administration of dabigatran, rivaroxaban, apixaban, or edoxaban
- Chronic anticoagulation: Patients receiving chronic oral anticoagulation regardless findings at continuous electrocardiographic monitoring
  Interventions: Drug: Chronic administration of dabigatran, rivaroxaban, apixaban, or edoxaban

INTERVENTIONS:
Drug: Intermittent administration of dabigatran, rivaroxaban, apixaban, or edoxaban — Patients will receive intermittent treatment with a novel oral anticoagulant drug
  Other Names: INTERMITTENT GROUP
  Groups: Intermittent anticoagulation
Drug: Chronic administration of dabigatran, rivaroxaban, apixaban, or edoxaban — Patients will receive chronic treatment with a novel oral anticoagulant drug
  Other Names: CHRONIC GROUP
  Groups: Chronic anticoagulation

SUMMARY:
Preliminary experiences suggest that intermittent anticoagulation guided by continuous electrocardiographic monitoring can reduce the incidence of bleeding in patients with episodes of atrial fibrillation.

Uncertainty about the potential implications of a strategy of intermittent anticoagulation after percutaneous coronary intervention exists.

The investigators will perform a case-control study to evaluate the safety and efficacy of anticoagulation on demand in high bleeding risk (HBR) patients with paroxysmal atrial fibrillation after percutaneous coronary intervention.

DETAILED DESCRIPTION:
For decades now, stroke prevention in patients with atrial fibrillation has largely consisted of chronic oral anticoagulation, often with no end in sight. This strategy, however, is associate with a high incidence of bleeding complications, especially when anticoagulation is associated with antiplatelet agents, as it occurs in patients with coronary artery disease undergoing percutaneous coronary intervention.

Known as intermittent, on demand, or 'pill in the pocket' anticoagulation, the strategy of prescribing oral anticoagulation only when is actually needed, has gotten a feasibility boost from recent advancements in both medical therapy and rhythm monitoring technology.

Preliminary experiences suggest that intermittent anticoagulation guided by continuous electrocardiographic monitoring can reduce the incidence of bleeding in patients with episodes of atrial fibrillation.

Uncertainty about the potential implications of a strategy of intermittent anticoagulation after percutaneous coronary intervention exists.

The investigators will perform a case-control study to evaluate the safety and efficacy of anticoagulation on demand in high bleeding risk (HBR) patients with paroxysmal atrial fibrillation after percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* No chronic atrial fibrillation
* Coronary artery disease
* Percutaneous coronary intervention

Exclusion Criteria:

* Contraindications to anticoagulation
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High bleeding risk (HBR) patients undergoing percutaneous coronary angiography with history of paroxysmal atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Outcome Event (MACE) | Up to 1 year
  The time to final occurrence of cardiovascular death, non-fatal myocardial infarction, ischemic stroke or ischemia driven revascularization
Days on anticoagulant treatment | Up to 1 year
  The total number of days on anticoagulant treatment

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Gaudio, MD, Study Director — University Sapienza
Locations (2):
- Italy (2):
  - San Raffaele Pisana, Rome
  - Sapienza University, Rome

IPD SHARING:
Plan to Share IPD: Undecided